CLINICAL TRIAL: NCT06385782
Title: Reduce of Heart Rate Variability of Asian Antarctic Overwintering Members and the Impact Factors--A Prospective Observational Study
Brief Title: Exploring HRV in Antarctic Overwintering Members of Asia
Status: Completed | Type: Observational
Sponsor: Ya-Wei Xu (Other)
Responsible Party: Sponsor-Investigator, Ya-Wei Xu, PHD, Shanghai 10th People's Hospital
Organization: Shanghai 10th People's Hospital (Other)
Other Study IDs: 20dz1207200
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Heart Rate Variability
Keywords: Heart Rate Variability (HRV); Antarctic Regions; Overwintering; Physical harm; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- outdoor groups: Outdoor work time is more than 2 hours
  Interventions: Other: Antarctic environment
- indoor groups: Outdoor work time is less than 2 hours
  Interventions: Other: Antarctic environment

INTERVENTIONS:
Other: Antarctic environment — . According to the different work content of the scientific expedition team members, and taking the average outdoor working time of 2 hours/day as the node, the scientific expedition team members are divided into outdoor groups (n=12) and indoor groups (n=10). Participants will be assessed on the day they enter the Antarctic station and leave.

SUMMARY:
Extreme changes in the Antarctic environment can cause emotional and autonomic dysfunction. In this study, volunteers from the Antarctica stations in China provided scale scores and heart rate variability (HRV) data, which were used to assess the autonomic nervous system. Enroll twenty-two members from Zhongshan Station and the Great Wall Station who are overwintering. Using the Generalized Anxiety Disorder (GAD-7) scale, the Patient Health Questionnaire-9 (PHQ-9) scale, and the SF-36 quality of life scale to evaluate the individual's general physical and mental health. Analyze HRV and other associated parameters.

DETAILED DESCRIPTION:
This study was a prospective observational study. We selected 12 members in Antarctica at the Great Wall Station of the 37th Chinese Antarctic Scientific Expedition (CSEA) from March 2021 to April 2022. And 10 members in Antarctica at Zhongshan Station in the 38th CSEA from December 2021 to April 2023. There were 22 members in total. Team members are volunteers selected through interviews, followed by detailed medical and psychological examinations, and are made up of scientific and logistical staff. According to the different work content of the scientific expedition team members, and taking the average outdoor working time of 2 hours/day as the node, the scientific expedition team members are divided into outdoor groups (n=12) and indoor groups (n=10). Participants will be assessed on the day they enter the Antarctic station and leave. Assessments include HRV, SF-36 quality of life questionnaire, Patient Health Questionnaire-9 (PHQ-9) scale and Generalized Anxiety Disorder (GAD-7) scale. This study approved by the local ethics committee of Shanghai Tenth People's Hospital, and conformed to the Declaration of Helsinki and its later amendments.

ELIGIBILITY:
Inclusion Criteria:

* Team members are volunteers selected through interviews, followed by detailed medical and psychological examinations, and are made up of scientific and logistical staff.

Exclusion Criteria:

* People with physical or mental illness

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study was a prospective observational study. We selected 12 members in Antarctica at the Great Wall Station of the 37th Chinese Antarctic Scientific Expedition (CSEA) from March 2021 to April 2022. And 10 members in Antarctica at Zhongshan Station in the 38th CSEA from December 2021 to April 2023. There were 22 members in total. Team members are volunteers selected through interviews, followed by detailed medical and psychological examinations, and are made up of scientific and logistical staff.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
changes in HRV | members in Antarctica at Zhongshan Station in the 38th CSEA from December 2021 to April 2023
  Before and after the expedition to Antarctica, we conducted comparative analyses of HRV data.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No